CLINICAL TRIAL: NCT00162474
Title: Correlation Between Phenotypic Activity of CYP2C9 and Genetic Polymorphism in CYP2C9 and Warfarin Metabolism.
Brief Title: Determinants of Warfarin Metabolism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: yc195510-HMO-CTIL
Record Dates: First submitted 2005-09-11; First posted 2005-09-13 (Estimated); Last update posted 2018-06-12 (Actual); Status verified 2018-03

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — Warfarin; Phenytoin

ARMS (1):
- Warfarin (Experimental)
  Interventions: Drug: Warfarin; Drug: Phenytoin

INTERVENTIONS:
Drug: Warfarin
Drug: Phenytoin

SUMMARY:
The anticoagulant effect of warfarin varies greatly among individuals. Some of this variability is attributed to differences in the activity of CYP2C9, the predominant enzyme involved in the metabolism of S-warfarin.

The present study is designed to define the differences in warfarin metabolism among healthy individuals carrying different CYP2C9 genotypes. In addition, the study will define the correlation between the phenytoin metabolic ratio, a marker of CYP2C9 activity in vivo, and warfarin metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Age range of 20-50 years old
* The absence of significant disease states

Exclusion Criteria:

* Known hypersensitivity to warfarin or phenytoin
* The presence of significant disease states
* Regular use of drugs (including birth control pills)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2003-09; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Warfarin oral clearance | 2 weeks
Formation clearance of CYP2C9 mediated warfarin metabolites | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Caraco, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel

REFERENCES:
- [Derived] Shaul C, Blotnick S, Muszkat M, Bialer M, Caraco Y. Quantitative Assessment of CYP2C9 Genetic Polymorphisms Effect on the Oral Clearance of S-Warfarin in Healthy Subjects. Mol Diagn Ther. 2017 Feb;21(1):75-83. doi: 10.1007/s40291-016-0247-7. PMID 27878474